CLINICAL TRIAL: NCT02807792
Title: Perianal Operating Scope Feasibility
Brief Title: Perianal Operating Scope Feasibliity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1601M83061
Record Dates: First submitted 2016-05-18; First posted 2016-06-21 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Transanal Endoscopic Surgery
Keywords: Perianal surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Perianal access device (Experimental)
  Interventions: Device: Perianal access device

INTERVENTIONS:
Device: Perianal access device — Perianal access device

SUMMARY:
This protocol will test a new prototype of a peri-anal access device, with increased flexible length and a captured operative field, for feasibility in patients immediately prior to their scheduled peri-anal procedure.

DETAILED DESCRIPTION:
Research Methods: The insertion of the modified access device in five patients before their planned peri-anal procedure, which will subsequently be performed with standard instruments, will allow us to observe the ease of insertion, the expansion of the blades, and the creation of the operative field achieved. If necessary, we will modify our design based on these findings. When a successful, operating room prototype is established, the device will be suitable for clinical use and the stated benefits thereof.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 to 80
* In good health status
* Patients scheduled for a transanal procedure other than for anal lesions, e.g., hemorrhoids, fissures, abscesses

Exclusion Criteria:

* Patients with physical characteristics that distort the rectal sigmoid anatomy, e.g., spinal lesions.
* Patients considerable unsuitable for inclusion in the study by their colorectal surgeon.
* Patients considered too frail or ill by their physician to undergo a 5-10 minute prolongation of their procedure.
* Patients with known rectosigmoid infections.
* Patients with known rectosigmoid wall fragility.
* Patients with known rectosigmoid perforations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Visual assessment of operative field dimensions measured in centimeters | Baseline
  The Outcome Measure Title implies the visual measurement that will be used to describe the potential operative field delineated by our experimental perianal access device. The description will, therefore, be primarily a qualitative visual assessment with the addition of estimated dimensions measured in centimeters for the length of the longitudinal and transverse fields encompassed by the blades of the access device. The collected measurement data will be aggregated, the numerical data averaged, and the visual perceptions integrated. The Time Frame for the individual study of each insertion will be two minutes or less. There is no chronic component to this feasibility analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Buchwald, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided